CLINICAL TRIAL: NCT06161402
Title: The Effectiveness of an Elastic Band -Based Progressive Resistance Training (EB-PRT) in Improving Sarcopenia and Clinical Outcomes Among Patients With Heart Failure: A Pilot Mixed-method Study
Brief Title: Elastic Band-Progressive Resistance Training (EB-PRT) for Sarcopenia Among Heart Failure Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EB-PRT
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Sarcopenia; Resistant Training
MeSH Terms: conditions — Heart Failure; Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EB-PRT (Experimental): EB-PRT will implemented during week 1-14. A purposive sample of 12 participants invited for qualitative interview during 21st -22nd week. There are 2 post-test evaluations at 14th week and 26th week. After the second evaluation at week 26, the group will receive usual care with routine follow-up.
  Interventions: Behavioral: Elastic band-based progressive resistance training (EB-PRT)
- Usual care (No Intervention): The control group will receive usual care including the medical care offered by the specialist out-patient clinic during 1-26 week. There are 2 post-test evaluations at 14th week and 26th week. From week 27 to week 40, this wait-list control group will receive the same EB-PRT as the intervention group.

INTERVENTIONS:
Behavioral: Elastic band-based progressive resistance training (EB-PRT) — EB-PRT will be implemented during week 1-14. The EB-PRT comprises a 4-week training phase, 6-week consolidation phase and a 4-week maintenance phase.
  Arms: EB-PRT

SUMMARY:
Heart failure (HF) is a complicated clinical syndrome caused by structural and/or functional cardiac abnormalities that result in ineffective myocardial pumping. HF management has placed more emphasis on improving the prognostic factors which determine these poor clinical outcomes. More recently, the prognostic role of sarcopenia in HF has received particular attention. Defined as progressive and generalized decline in skeletal muscle mass, strength and physical performance due to aging, sarcopenia is definitely a common comorbid of HF which follows an age-specific disease epidemiology. Given muscle disuse is the most preventable and reversible factor of sarcopenia, more evidence points to the therapeutic value of resistance training (RT) for this debilitating condition. Nevertheless, the therapeutic effects of RT on improving sarcopenia and thereby the disease prognosis among HF patients is yet to be evaluated. Therefore, the sequential mixed method study including a pilot RCT will be conducted to evaluate the preliminary effect of a 14-week elastic band-progressive resistance training (EB-PRT) and a subsequent qualitative study to explore the subjects' engagement experience. The outcomes cover the whole set of defining characteristics including muscle mass, muscle strength and functional performance and the clinical outcomes which reflect HF disease severity and patient-reported HRQL.

DETAILED DESCRIPTION:
The aim of this study is to investigate the therapeutic value of resistant training (RT) in improving sarcopenia in heart failure patients. To better achieve such therapeutic effects, the design of RT program also needs to comply with the exercise guideline with emphasis placed on increasing the skeletal muscle mass (i.e., the key pathological factor of sarcopenia). Addressing these research agenda is crucial to inform the development of evidence-based practice to tackle the prognostic impact of sarcopenia among HF patients. This is a sequential mixed method study including a pilot RCT to evaluate the preliminary effect of a 14-week elastic band-progressive resistance training (EB-PRT) and a subsequent qualitative study to explore the subjects' engagement experience. The total study period last for 40 weeks. The sample size is 62 participants. It is a single-blinded study. The research assistants for data collection will be blinded.

For intervention group, EB-PRT is implemented during week 1-14. A purposive sample of 12 participants invited for qualitative interview during 21st -22nd week. There are 2 post-test evaluations at 14th week (T1) and 26th week (T2). After the second evaluation at week 26, the group will receive usual care with routine follow-up. For the qualitative study on, a subsample of 12 participants in intervention group will be invited to explore their experience and perception at about 21st-22th week. The interview will be semi-structured and taken about 30-40 minutes at participants' home. The control group will receive usual care including the medical care offered by the specialist out-patient clinic during 1-26 week. There are 2 post-test evaluations at 14th week (T1) and 26th week (T2). From week 27 to week 40, this wait-list control group will receive the same EB-PRT as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 50;
2. has a confirmed clinical diagnosis of HF in the electronic health record for at least 6 months to ensure adequate disease exposure;
3. meeting the Asian Working Group of Sarcopenia's criteria2 [grip strength measured by dynamometer (Male: <28kg; Female: <18kg); low physical function (defined by Short Physical Performance Battery score ≤9) and reduced muscle mass by bioimpedance analysis (Inbody Technology 270; Male: appendicular skeletal muscular index (ASMI) <7.0kg/m2, Female: <5.7kg/m2)];
4. has stable HF and do not have any acute respiratory and musculo-skeletal condition which contradict them from practising exercise;
5. no regular resistance training for the previous 6 months.

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Appendicular skeletal muscular index (ASMI) | Changes from baseline to 14 weeks (1st post-test) and 26 weeks (2nd post-test).
  ASMI will be measured by the bioimpedance analysis (BIA) method. Reduced muscle mass is defined if ASMI <7.0kg/m2 for male, ASMI <5.7kg/m2 for female.
Handgrip strength | Changes from baseline to 14 weeks (1st post-test) and 26 weeks (2nd post-test).
  Handgrip strength will be measured by a hydraulic hand dynamometer from dominant hand, taking the highest value among 3 measurements. Low muscle strength is defined if male <28kg, and femal <18kg.
Physical function | Changes from baseline to 14 weeks (1st post-test) and 26 weeks (2nd post-test).
  Physical function will be measured by the Short Physical Performance Battery (SPPB), which combines balance test, gait velocity and chair stand. SPPB score ranges from 0-12, higher score better physical performance. Low physical function is defined by SPPB score ≤9.

SECONDARY OUTCOMES:
Symptom burden | Changes from baseline to 14 weeks (1st post-test) and 26 weeks (2nd post-test).
  Symptom burden will be measured by the Memorial Symptom Assessment Scale (MSAS-HF). The total symptom scores are summed to obtain a final grand total symptom burden score (score range of 0 to 416). Higher scores indicate greater symptom burden.
Health-Related Quality of Life (HRQL) | Changes from baseline to 14 weeks (1st post-test) and 26 weeks (2nd post-test).
  HRQL will be measured by the 21-item Minnesota Living with Heart Failure Questionnaire (MLHFQ), to capture the physical, emotional and social well-being. MLHFQ provides a total score (range 0-105, from best to worst HRQoL).

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided